CLINICAL TRIAL: NCT01394419
Title: Effect of N-acetylcysteine on Prevention of Acute Kidney Injury in High Risk Patients Undergoing Off-pump Coronary Artery Bypass Graft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2010-0135
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Postoperative Acute Kidney Injury After Off-pump Coronary Artery Bypass Graft
MeSH Terms: interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC group (Experimental): N-acetylcysteine
  Interventions: Drug: N-acetylcysteine
- Placebo group (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 150 mg/kg bolus over 15 min after induction of anesthesia, followed by an infusion of 150 mg/kg/day for 24 hrs
  Arms: NAC group
Drug: Saline — Equal volume of normal saline
  Arms: Placebo group

SUMMARY:
N-acetylcysteine may prevent acute kidney injury in high risk patients undergoing off-pump coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing off-pump coronary artery bypass surgery and meets more than one of the following criteria;

  * preoperative serum creatinine > 1.4 mg/dl
  * Age > 70 years
  * Diabetes mellitus
  * left ventricular ejection fraction < 35 % or congestive heart failure (NYHA III or IV)
  * emergency surgery or re-operation

Exclusion Criteria:

* preoperative acute renal failure, patients on dialysis, use of N-acetylcystein within 5 days of surgery, history of hypersensitivity to N-acetylcystein

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | within 5 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Song JW, Shim JK, Soh S, Jang J, Kwak YL. Double-blinded, randomized controlled trial of N-acetylcysteine for prevention of acute kidney injury in high risk patients undergoing off-pump coronary artery bypass. Nephrology (Carlton). 2015 Feb;20(2):96-102. doi: 10.1111/nep.12361. PMID 25384603